CLINICAL TRIAL: NCT06121856
Title: VerioVue Enhancements Regulatory Clinical Evaluation - Professional Comparison to Validated Method: Arterial Study
Brief Title: Project VerioVue Enhancements - Arterial Study
Status: Completed | Type: Observational
Sponsor: LifeScan Scotland Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: FILE-PROT-005439
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- In-patients cardiothoracic intensive care: In-patients in the cardiothoracic intensive care department that were at least 16 years old and were fitted with an arterial line. There was no requirement to have diabetes but the study aimed to recruit a minimum of 20% subjects with diabetes.
  Interventions: Device: VerioVue Enhancements BGMS

INTERVENTIONS:
Device: VerioVue Enhancements BGMS — Blood glucose monitoring system

SUMMARY:
The aim of this performance evaluation is to compare the blood glucose results obtained using the VerioVue Blood Glucose Monitoring System (BGMS) with those obtained from a validated comparator method (iSTAT 1 Analyser) using arterial blood. The main question the study aims to answer is:

How accurate is the VerioVue BGMS when compared to a product that has already been confirmed as accurate (iSTAT 1 Analyser) when hospital staff test arterial blood on these two types of instrument? Participants will have a small amount of blood taken from an existing arterial line.

DETAILED DESCRIPTION:
Up to two UK NHS hospital sites will be used to collect a minimum of 100 evaluable samples from participants fitted with an arterial line that meet the acceptance criteria. Consent will be obtained from the participants prior to taking part in the study. If the participant meets the enrolment criteria then demographics and medical history information will be collected. A small volume of blood (max 150µl) will be collected from an existing arterial line. The blood will then be applied to six investigational OneTouch VerioVue meters (with expanded haematocrit range 20-65%) fitted with OneTouch Verio test strips and the blood glucose meter readings recorded. Three different lots of test strips will be used in rotation across the study. Within 5 minutes of the last meter test, trained staff will use blood from the same sample and perform a test on the iSTAT Analyser to obtain the blood glucose, haematocrit and oxygen levels of the sample. No treatment decisions will be made based on the blood glucose results obtained for this study. The study documentation will be reviewed by LifeScan monitors for completeness and accuracy and the results entered into a validated database. The data will be extracted and statistically analysed to determine the accuracy of the arterial blood glucose results obtained using the OneTouch VerioVue BGMS when compared to the arterial blood glucose results obtained on the iSTAT 1 Analyser.

ELIGIBILITY:
Inclusion Criteria:

Age - The potential Subject is at least 16 years old. Language - Subject reads and understands English. Informed Consent - The potential subject must read the Participant Information Sheet and sign the Informed Consent Form.

Subject agrees to provide relevant demographic, medical history, and prescription medication information.

The subject agrees to allow study staff access to medical records where necessary.

The Subject agrees to all aspects of the study process, including arterial blood draws performed by an HCP.

Exclusion Criteria:

Age - Subject is under 16 years old. Current Covid-19 positive test result.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will comprise a minimum of 100 evaluable samples taken from participants who are in the cardiothoracic intensive care unit of an NHS hospital who have an arterial line fitted for other medical purposes.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Performance evaluation: blood glucose monitoring system accuracy: BGMS vs reference instrument using arterial blood | Within 30 minutes of arterial blood sample draw.
  Performance Evaluation to compare the VerioVue BGMS blood glucose results to results obtained using the iSTAT 1 Analyser, a validated comparator method when using arterial blood.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Zammitt, MBChB, Principal Investigator — Edinburgh Centre for Endocrinology and Diabetes
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No